CLINICAL TRIAL: NCT01934231
Title: A Multicenter, Open-Label Study To Assess The Efficacy And Safety Of Potassium Clavulanate/Amoxicillin (CVA/AMPC 1:14 Combination) In The Treatment Of Children With Acute Bacterial Rhinosinusitis
Brief Title: Study to Assess the Efficacy and Safety of Potassium Clavulanate/Amoxicillin in Children With Acute Bacterial Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117150
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Sinusitis, Acute
Keywords: Acute bacterial rhinosinusitis; Amoxicilin; Infection; Potassium clavulanate
MeSH Terms: conditions — Sinusitis; Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Each participant will take Potassium Clavulanate (CVA)/ Amoxicillin (AMPC) corresponding 6.4/90 mg/kg/day in two divided doses (every 12 hours) just before lactation or meal for 7 days depending on his/her body weight at the start of treatment (Day 1). The actual daily dose depends on the body weight of the participant.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate Combination — The drug is available in two sachets (CVA/AMPC Dry Syrup 0.505 g and CVA/AMPC Dry Syrup 1.01 g). CVA/AMPC Dry Syrup 1.01 g sachet contains 42.9 mg of Potassium Clavulanate and 600 mg of Amoxicillin Hydrate. It is a white to yellowish white powder and has strawberry flavor and it is white to yellowish white suspension when it is suspended before use.

SUMMARY:
Acute Bacterial Rhinosinusitis (ABRS) is a respiratory inflammation commonly seen in clinical practice, which has with respiratory symptoms including nasal congestion, rhinorrhoea, postnasal discharge and cough and is associated with headache, cheek pain, facial pressure and other conditions. The principal bacterial pathogens in causing ABRS include Streptococcus pneumoniae, Haemophilus influenzae and Moraxella (Branhamella) catarrhalis. These three bacteria account for approximately 90% of ABRS in children less than or equal to 5 years of age. Combination of Potassium Clavulanate (CVA) and Amoxicillin (AMPC) produces higher antibiotic activity against beta-lactamase-producing bacteria. The present study is designed to assess the clinical efficacy, bacteriological efficacy and safety of CVA/AMPC (1:14) administered in children aged from 3 months to less than 15 years with ABRS. It is an open-label study consisting of a 7-day treatment phase and a post-treatment follow-up phase for 7 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Child with ABRS with inflammation as bacterial infection who has the following symptoms/signs on the day of or the day before the first dose of the investigational product: Redness of the nasal mucosa; nasal or postnasal discharge is purulent or mucopurulent; Pathological shadow in the paranasal sinus on a radiogram (only for reference). Patient with surgical history should be excluded but patient with a pervious surgery more than 365 days before and apparently preserved maxillary sinus mucosa or patient with a previous surgery of nasal polypectomy more than 90 days before may be enrolled in the study.
* Child with ABRS whose severity is classified as moderate or severe (total score >=4) based on the nasal cavity findings and symptoms.
* Boy or girl aged >=3 months to <15 years.
* Body weight >=6 kilograms (kg) to <40 kg.
* Written informed consent has been obtained from the child's legally acceptable representative. If the child is 12 years or older, the child him/herself should have also provided written informed consent. The investigator (or sub-investigator) should attempt to obtain written informed consent from the child him/herself as far as possible even if the child is less than 12 years of age.

Exclusion Criteria:

* Severe infection that requires surgical treatment (e.g., child with systemic symptoms such as fever associated with swelling face, child with almost full nasal obstruction due to a large nasal polyp).
* Serious complication such as acute mastoiditis, facial palsy, bacterial meningitis, and brain tumor.
* Congenital disorder such as maxillofacial dysplasia.
* Need of concomitant use of other antibiotics.
* Serious underlying disease (e.g., cardiac disease, malignancy, juvenile diabetes).
* Concurrent infection associated with gastrointestinal symptoms (e.g., diarrhoea, vomiting) that may affect safety assessment.
* Known hypersensitivity to any component of CVA/AMPC or penicillin or cephem antibiotic, or past history of a serious adverse reaction possibly related to any of these agents.
* Infectious mononucleosis.
* Current hepatic impairment, or past history of jaundice or hepatic impairment due to any component of CVA/AMPC.
* Past or current renal impairment (e.g., serum creatinine >=1.5 × Upper Limit of Normal, creatinine clearance of less than 30 milliliter/liter [mL/L]).
* Past or current immune dysfunction or insufficiency, or use of immunosuppressive therapy.
* Need corticosteroid for systemic, eye drops or nasal drops.
* Phenylketonuria.
* Use of azithromycin within 14 days prior to the first dose of the investigational product.
* Use of any antibiotic within 7 days prior to the first dose of the investigational product.
* Current use or imperative use during the study period of probenecid or a tubular secretion inhibitor.
* Participation in another clinical study within 3 months prior to enrollment, or prospected participation in another clinical study during the period of this study.
* Girl with menstruation and childbearing potential, pregnant girl, lactating girl, or girl who is planning a pregnancy during the study period. A girl with childbearing potential may be enrolled in the study only if she is willing to use at least one of the following acceptable measures for contraception throughout the study period: Male partner sterilization prior to the girl's entry into the study, and this male is the sole partner for that girl; Intrauterine device (IUD) (with documented annual failure rate estimate of <1%); Abstinence; Male condom combined with a female diaphragm, either with or without a vaginal spermicide.
* The legally acceptable representative is a minor.
* Child in care.
* History of alcohol or drug abuse.
* Relationship with the study medical institution: The investigator, sub-investigator, study collaborator, person employed by the investigator or the study medical institution, or their close relatives.
* Child whose participation in the study is considered inappropriate by the investigator (or sub-investigator).

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2013-11-07 (Actual); Study Completion 2013-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117150 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- CVA/AMPC (1:14): Participants received an oral dose of dry syrup potassium clavulanate (CVA)/amoxicillin hydrate (APMC) for 7 days. The daily dose of CVA/AMPC (1:14) was equal to CVA 6.4 milligrams (mg) (potency)/kilogram (kg)/day and AMPC 90 mg (potency)/kg/day in two divided doses (every 12 hours) just before lactation or meal depending on body weight at the start of treatment (Day 1).
Period: Overall Study
Arm/Group | CVA/AMPC (1:14)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Outcome of "Cure" at Test of Cure (TOC: Day 15)
Description: Clinical assessment of acute bacterial rhinosinusitis was performed by the investigator (or subinvestigator) at TOC (Day 15) on the basis of the following criteria: "Cure" is defined as sufficient resolution or improvement of the signs and symptoms such that no additional antibiotic therapy is needed. Failure is defined as no change or deterioration of the signs and symptoms or as additional antibiotic therapy being needed. The outcome was unable to be determined if no information was available regarding the signs and symptoms or, despite improvement of the signs and symptoms, the use of a non-study antibiotic was administered, indicating that there was a protocol deviation.
Time Frame: Day 15
Population: Per Protocol (PP) Population: all participants randomized to treatment who received the study drug for at least the first 3 days of study treatment in the Treatment Period and had evaluable data on both Day 8 and Day 15 with treatment compliance between 80% and 100% and no major protocol deviations
Measure: Number; unit: Participants
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 26
Participants
  Cure | 23
  Failure | 3
  Unable to Determine | 0
Statistical Analysis 1: Comparison: CVA/AMPC (1:14); Test type: Superiority or Other; Rate of Cure = 88.5, 95% CI 2-sided [69.85 to 97.55] — The estimated parameter represents the rate of cure, calculated as (number of participants with an outcome of "Cure"/number of participants analyzed) * 100

2. Secondary Outcome: Number of Participants With a Clinical Outcome of "Cure" at the End of Treatment (EOT: Day 8)
Description: Clinical assessment of acute bacterial rhinosinusitis was performed by the investigator (or subinvestigator) at the EOT (Day 8) on the basis of the following criteria: "Cure" is defined as sufficient resolution or improvement of the signs and symptoms such that no additional antibiotic therapy is needed. Failure is defined as no change or deterioration of the signs and symptoms or as additional antibiotic therapy being needed. The outcome was unable to be determined if no information was available regarding the signs and symptoms or, despite improvement of the signs and symptoms, the use of a non-study antibiotic was administered, indicating that there was a protocol deviation.
Time Frame: Day 8
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 26
Participants
  Cure | 25
  Failure | 1
  Unable to Determine | 0

3. Secondary Outcome: Number of Participants With a Clinical Outcome of "Cure" at Both the End of Treatment and Test of Cure (EOT and TOC: Day 8 and Day 15)
Description: Clinical assessment of acute bacterial rhinosinusitis was performed by the investigator (or subinvestigator) at the EOT (Day 8) and TOC (Day 15) on the basis of the following criteria: "Cure" is defined as sufficient resolution or improvement of the signs and symptoms such that no additional antibiotic therapy is needed. Failure is defined as no change or deterioration of the signs and symptoms or as additional antibiotic therapy being needed. The outcome was unable to be determined if no information was available regarding the signs and symptoms or, despite improvement of the signs and symptoms, the use of a non-study antibiotic was administered, indicating that there was a protocol deviation. In order to be categorized as "cure," participants had to meet the criteria for "cure" at both Day 8 and Day 15.
Time Frame: Day 8 and Day 15
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 26
Participants
  Cure | 23
  Failure | 3
  Unable to Determine | 0

4. Secondary Outcome: Number of Participants With the Indicated Severity of Symptoms and Nasal Cavity Findings at Day 4, Day 8, and Day 15
Description: The investigator (or sub-investigator) categorized the severity of symptoms such as rhinorrhoea and bad mood/productive cough as none, mild/small amount (M/SA), or moderate or severe (M or S). For the nasal cavity finding of nasal/postnasal discharge (N/PD) the categozation was serous [containing serum]), mucopurulent (MU/SA [containing both mucus and pus]), and moderate or larger amount (M/LA). In cases in which both sides of the nasal cavity were affected and there was no difference in severity between the sides, the right-side results were recorded. If there was a difference in severity, the more severe-side results were recorded.
Time Frame: Baseline (BL), Day 4, Day 8, and Day 15
Population: PP Population
Measure: Number; unit: Participants
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 26
Participants
  Rhinorrhoea: BL, None | 0
  Rhinorrhoea: BL, M/SA | 5
  Rhinorrhoea: BL, M or S | 21
  Rhinorrhoea: Day 4, None | 7
  Rhinorrhoea: Day 4, M/SA | 16
  Rhinorrhoea: Day 4, M or S | 3
  Rhinorrhoea: Day 8, None | 13
  Rhinorrhoea: Day 8, M/SA | 13
  Rhinorrhoea: Day 8, M or S | 0
  Rhinorrhoea: Day 15, None | 18
  Rhinorrhoea: Day 15, M/SA | 8
  Rhinorrhoea: Day 15, M or S | 0
  Bad mood/productive cough: BL None | 4
  Bad mood/productive cough: BL, M/SA | 20
  Bad mood/productive cough: BL, M or S | 2
  Bad mood/productive cough: Day 4, None | 16
  Bad mood/productive cough: Day 4, M/SA | 10
  Bad mood/productive cough: Day 4, M or S | 0
  Bad mood/productive cough: Day 8, None | 21
  Bad mood/productive cough: Day 8, M/SA | 5
  Bad mood/productive cough: Day 8, M or S | 0
  Bad mood/productive cough: Day 15, None | 24
  Bad mood/productive cough: Day 15, M/SA | 2
  Bad mood/productive cough: Day 15, M or S | 0
  N/PD: BL, Serous | 0
  N/PD: BL, MU/SA | 6
  N/PD: BL, M/LA | 20
  N/PD: Day 4, Serous | 14
  N/PD: Day 4, MU/SA | 10
  N/PD: Day 4, M/LA | 2
  N/PD: Day 8, Serous | 22
  N/PD: Day 8, MU/SA | 4
  N/PD: Day 8, M/LA | 0
  N/PD: Day 15, Serous | 21
  N/PD: Day 15, MU/SA | 5
  N/PD: Day 15, M/LA | 0

5. Secondary Outcome: Number of Participants (Par.) With the Specified Bacteriological (Bact.) Outcome Per Pathogen (Path.) at the End of Treatment (EOT) at Day 8
Description: The investigator used the sample collected at the start of study treatment (trt) to isolate and identify the pathogenic bacteria. The sample collected at the EOT was used to evaluate the bact. response to the investigational product of each path. If the same pathogen was not detected at the EOT, this pathogen was classified as "eradication" (E). If the same pathogen was detected at the EOT, this pathogen was classified as "persistence" (P).
Time Frame: Day 8
Population: Bacteriology PP Population: all participants in the PP Population, excluding the participants who were classified as "Unable to determine" for the bacteriological outcome and who had no identified pathogen at Day 1
Measure: Number; unit: Participants
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 24
Participants
  Streptococcus pneumoniae (StPn), E | 8
  StPn, P | 1
  Penicillin Susceptible (PenSusc) StPn, E | 7
  PenSuscStPn, P | 1
  Pen Intermediate (PenInt) StPn, E | 1
  PenIntStPn, P | 0
  Pen Resistant (PenR) StPn, E | 0
  PenRStPn, P | 0
  Moraxella (Branhamella) catarrhalis (MBC), E | 6
  MBC, P | 0
  MBC beta-lactamase (BL) positive, E | 6
  MBC BL positive, P | 0
  MBC BL negative (N), E | 0
  MBC BLN, P | 0
  Haemophilus influenzae (HI), E | 8
  HI, P | 6
  HI BLN ampicillin (A) susceptible (S), E | 8
  HI BLNAS, P | 2
  HI BLNA resistant (R), E | 0
  HI BLNAR, P | 3
  HI BL Producing (Pr) AR, E | 0
  HI BLPrAR, P | 1
  Staphylococcus aureus (Staph Ar), E | 5
  Staph Ar, P | 0
  Methicillin R Staph Ar, E | 0
  Methicillin R Staph Ar, P | 0
  Streptococcus pyogenes, E | 1
  Streptococcus pyogenes, P | 0
  Enterobacter species (sp), E | 1
  Enterobacter sp., P | 0
  Coagulase (Coag) NStaph, E | 3
  CoagNStaph, P | 0
  Corynebacterium sp., E | 1
  Corynebacterium sp., P | 0
  Streptococcus sp., E | 1
  Streptococcus sp., P | 0
  Pseudomonas aeruginosa, E | 0
  Pseudomonas aeruginosa, P | 0

6. Secondary Outcome: Number of Participants (Par.) With the Specified Bacteriological (Bact.) Outcome Per Participant at EOT (Day 8)
Description: The investigator used the sample collected at the start of study treatment (trt) to isolate and identify the pathogenic bacteria. The sample collected at the EOT was used to evaluate the bact. response to the investigational product of each par. using the following classification: Bact. eradication (erad.), presumed bact. erad. and colonization were categorized as erad. Bact. persistence (pers.), presumed bact. pers. and superinfection were categorized as pers. Bact. erad. elimination of the pathogen (path.) after trt; presumed bact. erad.-resolution of signs/symptoms (s/s) after trt; colonization-resolution of s/s but initial path. still recovered from sample; bact. pers.-no improvement in s/s and initial path. was recovered from sample; presumed bact. pers.-no improvement in s/s and isolation of initial path. was impossible/not performed; superinfection-initial path. was eradicated but a new path. was recovered; unable to determine-bact. test could not be performed.
Time Frame: Day 8
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | CVA/AMPC (1:14)
Number analyzed (Participants) | 24
Participants
  Eradication | 24
  Persistence | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to Study Day 22).
Description: SAEs and non-serious AEs were reported for members of the Safety Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | CVA/AMPC (1:14)
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 5/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVA/AMPC (1:14) (N=27)
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Otitis media (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.